CLINICAL TRIAL: NCT04537325
Title: Prevention of Acute Kidney Injury After Transcatheter Aortic Valve Implantation in Patients With Chronic Kidney Disease With Controlled Intravenous Hydration Matched to Urinary Output
Brief Title: Prevention of Acute Kidney Injury After Transcatheter Aortic Valve Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AKI_TAVI
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Acute Kidney Injury
Keywords: Transcatheter aortic valve stenosis; Chronic kidney disease; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RenalGuard group (Active Comparator)
  Interventions: Device: RenalGuard system
- Control group (No Intervention)

INTERVENTIONS:
Device: RenalGuard system — Periprocedural intravenous hydration matched to urinary output.
  Arms: RenalGuard group

SUMMARY:
Randomized controlled, single-center trial randomizing patients with chronic kidney disease and symptomatic severe aortic valve stenosis undergoing transcatheter aortic valve implantation (TAVI). Patients are randomized in a 1:1 ratio to periprocedural intravenous hydration matched to urine output using the RenalGuard system and to standard hydration. The purpose of the study is to test, wether the controlled intravenous hydration with the RenalGuard system is superior to standard hydration to prevent acute kidney injury after TAVI.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) after transcatheter aortic valve implantation (TAVI) is associated with worse outcome. The RenalGuard system was developed to prevent AKI by a controlled furosemide-induced diuresis with matched isotonic intravenous hydration. It is based on the theory, that a high urinary output prevents contrast media-induced nephropathy (CIN).

The present study is a prospective, randomized trial to investigate wether a matched intravenous hydration using the RenalGuard system is superior to standard pre- and postprocedural intravenous hydration in patients with severe aortic valve stenosis and chronic kidney disease undergoing TAVI. Primary endpoint is the occurrence of AKI after TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic severe aortic valve stenosis undergoing transcatheter aortic valve implantation
* Chronic kidney disease (baseline glomerular filtration rate ≤ 60 ml/min)
* Written informed consent

Exclusion Criteria:

* Hemodynamic instability
* Dialysis-dependent chronic kidney injury
* Emergency transcatheter aortic valve stenosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | Within 7 days after Transcatheter aortic valve implantation
  Increase of serum-creatinine of 0,3 mg/dl in pre-procedural serum-creatinine within 7 days after Transcatheter aortic valve implantation

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schäfer, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Voigtlander-Buschmann L, Schafer S, Schmidt-Lauber C, Weimann J, Shenas M, Giraldo Cortes J, Kuta PM, Zeller T, Twerenbold R, Seiffert M, Schofer N, Schneeberger Y, Schafer A, Schirmer J, Reichenspurner H, Blankenberg S, Conradi L, Schafer U. Effect of periprocedural furosemide-induced diuresis with matched isotonic intravenous hydration in patients with chronic kidney disease undergoing transcatheter aortic valve implantation. Clin Res Cardiol. 2024 Jun;113(6):801-811. doi: 10.1007/s00392-023-02234-z. Epub 2023 Jun 1. PMID 37264143